CLINICAL TRIAL: NCT06917391
Title: The Young Adults' Experiences With Virtual Reality (YAES VR) Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 24-00910; 1K01MD019320-01A1 (NIH)
Record Dates: First submitted 2025-03-25; First posted 2025-04-08 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Population Health

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Reality (VR) food marketing exposure (Experimental): Participants will be given 15 minutes to explore the VR experience and provide feedback on whether they believe their peers would engage with the experience (concealment/deception).
  Interventions: Behavioral: Wendyverse VR food marketing experience
- VR non-food control (Active Comparator): Participants will be given 15 minutes to explore the VR experience and provide feedback on whether they believe their peers would engage with the experience (concealment/deception).
  Interventions: Behavioral: Nikeland VR non-food marketing experience

INTERVENTIONS:
Behavioral: Wendyverse VR food marketing experience — In the Wendyverse VR application ("app") participants can order from a Wendy's restaurant, play games, meet with others who may be visiting the Wendyverse, and access codes that can be used to obtain free food at physical restaurants.
  Arms: Virtual Reality (VR) food marketing exposure
Behavioral: Nikeland VR non-food marketing experience — In Nikeland VR app, participants can play sports, try on apparel, and engage with celebrity athletes.
  Arms: VR non-food control

SUMMARY:
The purpose of this study is to test the effect of virtual reality (VR) food marketing exposure (versus VR non-food control) on snack consumption, purchase intention, hunger, and arousal in black and white young adults. Participants will be randomized to either the VR food marketing condition or VR non-food control. Study participation duration will be 2 hours during a one-time, single visit.

DETAILED DESCRIPTION:
Food marketing has been unequivocally linked to poor diet and risk of excessive weight gain in young people. Food companies disproportionately target Black consumers with more advertisements ("ads") and the least healthy ads, contributing to nutritional disparities and nutrition-related diseases. To expand their reach, food companies have developed virtual reality (VR) marketing experiences that are engaging, highly sophisticated, and may more powerfully elicit biological signals precipitating a motivation to consume foods. Yet, little is known about how exposure to VR food marketing influences biological and behavioral outcomes among Black young adults. The interactional role of food/nutrition insecurity and exposure to VR food marketing among Black young adults is also unknown. There is a critical need to understand the biological and behavioral effects of VR food marketing among Black communities while the technology is in its infancy.

ELIGIBILITY:
Inclusion Criteria:

1. 18-24 years old;
2. self-identify as Black or white in order to determine racial/ethnic differences in responses to unhealthy VR-based food and beverage marketing;
3. self-report normal or corrected-to-normal vision from glasses or contacts;
4. self-report comfort and ability to walk around within a VR paradigm;
5. able to read, write, understand, and respond to all study materials (including the VR paradigm) in English
6. residing in the NYC-metropolitan area in order to be available for in-person study
7. capacity and willingness to provide consent

Exclusion Criteria:

1. report a history of disorders causing motion sickness or have a history of significant motion sickness, which could be triggered within the VR paradigm
2. self-report dietary restriction, such as food allergies or veganism, which may lead to different effects when exposed to food marketing;
3. Self-report disliking 50% or more of the snacks that will be offered during the laboratory test snack as determined by a score of 5 or less on the food preferences questionnaire, which may have a confounding effect on consumption;
4. report being pregnant or breastfeeding, which may affect hunger;
5. smoke or consume tobacco, which decreases salivary flow; or
6. self-report being very hungry based on 100 mm VAS hunger rating, which minimizes the burden to participants to fast prior to the visit and maximizes the ability to detect differences between groups.Those excluded for being very hungry will have the option of returning to the visit on a different day.

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-11-13 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Snack consumption | Post-VR exposure (up to 20 minutes)
  Following the VR exposure, snacks (health and unhealthy snacks) will be offered to participants with the instruction to eat ad libitum for 20 minutes. Snack consumption will be measured using a Cardinal Detecto stainless steel scale which transmits weight information wirelessly.
Purchase intention via self-report questionnaire | Post-VR exposure (~5-10 minutes)
  Purchase intention will be assessed using a self-report questionnaire. Questions include: How likely are you to buy food from any fast-food restaurant in the next 2 weeks? Scores will range from 0 ("Not at all") to 5 ("Highly likely"). Higher scores indicate a higher likelihood to purchase food from the restaurant.
Change in salivary flow | Baseline, post-VR exposure (~5-10 minutes)
  A dental roll will be placed horizontally under participants' tongues for 30 seconds pre- and post-VR exposure. Salivation will not be collected during the exposure so as not to disrupt the immersion. An increase in salivary flow indicates hunger.
Change in electrodermal activity | From baseline to post-VR exposure, up to 15 minutes
  Electrodermal activity refers to the changes in the electrical properties of the skin due to sweat secretion. Electrodermal activity is measured through skin conductance, two Ag-AgCl electrodes will be taped to the distal phalanx of the index and ring fingers on the participants' non-dominant hand. Electrodermal activity will be measured. A stronger electrodermal response indicates arousal.

CONTACTS AND LOCATIONS:
Overall Officials: Omni Cassidy, Ph.D., Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices) will be made available as soon as possible or at the time of associated publication. All data will be shared by the close of the award. Data will be made available, at minimum, for seven years. Upon reasonable request The investigator who proposed to use the data. Data are available for 5 years at a third party website (Open Science Framework: https://osf.io/).
Supporting Information: Study Protocol, SAP
Time Frame: Data will be made available as soon as possible or at the time of associated publication. All data to be shared will be shared by the close of the award. Data will be made available, at minimum, for seven years.
Access Criteria: Data are available for 5 years at a third party website (Open Science Framework: https://osf.io/).
URL: https://osf.io/

REFERENCES:
- [Derived] Cassidy O, Boyland E, Persky S, Troxel AB, Elbel B. Examining the Effect of Virtual Reality-Based Fast-Food Marketing on Eating-Related Outcomes in Young Adults: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2025 Sep 22;14:e69096. doi: 10.2196/69096. PMID 40982800